CLINICAL TRIAL: NCT03311360
Title: Chinese Society of Interventional Radiology
Brief Title: Drug Coated Balloon Versus Stenting in Patients With Symptomatic Vertebral Artery Stenosis：an Observational Clinical Study
Status: Completed | Type: Observational
Sponsor: Chinese Society of Interventional Radiology (Other)
Responsible Party: Sponsor
Other Study IDs: CSIR01
Record Dates: First submitted 2017-10-09; First posted 2017-10-17 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2019-01

CONDITIONS: Vertebral Artery Origin Stenosis
Keywords: vertebral artery origin stenosis; drug-coated balloon; stenting; medical treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- drug-coated balloon: patients with vertebral artery origin stenosis treated with drug-coated balloons
  Interventions: Device: drug-coated balloon
- bare metal stent: patients with vertebral artery origin stenosis treated with bare metal stent
  Interventions: Device: bare metal stent

INTERVENTIONS:
Device: drug-coated balloon — Orchid and Dahlia DCB
  Groups: drug-coated balloon
Device: bare metal stent — any type of bare metal stent
  Groups: bare metal stent

SUMMARY:
There are two arms in our trial, DCB group, BMS group.The investigators are going to investigate the safety and efficacy of all groups at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 80 years old;
2. TIA or non-disabling ischaemic stroke of the posterior circulation;
3. symptoms occurred in the 14 days and could not be relieved after 2 months of regular medication
4. stenosis of the vertebral artery of 50% or greater, diagnosed by both CT angiography or angiography;
5. NIHSS≤ 6;
6. score on the modified Rankin scale ≤ 3.

Exclusion Criteria:

1. Active bleeding or coagulation disorders or severe renal/liver impairment
2. allergy to iodinated contrast agent or related medicines;
3. acute stroke in 3 weeks
4. more than 1 stenosis at the target vessel or Distal vascular dysplasia (diameter≤3mm)
5. a potential cause of stenosis other than atherosclerosis
6. Severe stenosis was found in the anterior circulation artery(>70%)
7. intracranial hemorrhage or hemorrhagic stroke, intracranial tumor, cerebral arteriovenous malformation, or intracranial aneurysm in 30 days;
8. ISR patients;
9. Severe calcification lesion；
10. obvious thrombosis in vessel;
11. pregnancy;
12. a potential cause of TIA or minor stroke other than stenosis in a vertebral artery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients meet all of the inclusion criteria and none of the excusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of vascular death,non-fatal myocardial and non-fatal stroke in 12 months | 12 months
  vascular death,non-fatal myocardial and non-fatal stroke diagnosed by specialist physician

SECONDARY OUTCOMES:
lumen loss at 6 months | 6 months
  lumen loss measured by doppler untrasound
lumen loss at 12 months | 12 months
  lumen loss measured by doppler untrasound
restenosis at 6 months | 6 months
  restenosis was assessed by doppler untrasound
restenosis at 12 months | 12 months
  restenosis was assessed by doppler untrasound
traget lesion revascularizition at 12 months | 12 months
  traget lesion revascularizition including envascular intervention and Surgery
Incidence of safety events including vascular death,non-fatal myocardial infarction, or non-fatal stroke in 30 days | 30 days
  safety events including vascular death,non-fatal myocardial infarction, or non-fatal stroke diagnosed by investigators within 30 days after start of the treatment
stent fracture rate at 12 months | 12 months
  stent fracture was assessed by DSA

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Anzhen hospital, Beijing
  - The rockets army general hospital, Beijing
  - The first affiliated hospital of Dalian medical university, Dalian
  - The first affiliated hospital of Harbin medical university, Harbin
  - The first hospital of Jilin university, Jilin
  - Shengjing Hosptal of china medical university, Shenyang
  - Henan provincial peoples hospital, Zhengzhou
  - The first hospital of zhengzhou university, Zhengzhou
  - Zhengzhou center hospital, Zhengzhou